CLINICAL TRIAL: NCT01406379
Title: Comparison of Clip and Detachable Snare in Preventing Postpolypectomy Bleeding for Pedunculated Colonic Polyps: a Prospective, Randomized Study
Brief Title: Comparison of Prophylactic Clip and Detachable Snare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong-Seon Ji, MD, PhD, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prophylatic clip
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic clip (Experimental): Prophylactic clip
  Interventions: Procedure: Prophylactic clip
- Detachable snare (Active Comparator): Detachable snare
  Interventions: Procedure: Detachable snare

INTERVENTIONS:
Procedure: Prophylactic clip — Before conventional snare polypectomy, hemoclips were applied on the base of stalk in the prophylactic clip group
  Arms: Prophylactic clip
Procedure: Detachable snare — In the detachable snare group, detachable snare was positioned at the base of stalk and followed by conventional snare polypectomy
  Arms: Detachable snare

SUMMARY:
Although endoscopic colonic polypectomy has been an established procedure for two decades, the risk of bleeding is still higher after resecting of pedunculated polyps, because of the presence of a large artery in the stalk. Several preventive methods such as detachable snare and adrenaline injection have been proposed in the management of postpolypectomy bleeding in large colonic polyps. For prophylactic clip, there was no prospective randomized study assessing the efficacy in the prevention of postpolypectomy bleeding for the large pedunculated polyps. So we designed a prospective, randomized study to compares the efficacy of application of prophylactic clip and detachable snare in the prevention of postpolypectomy bleeding in large polyps. Application of prophylactic clip will be as effective and safe method as detachable snare in the prevention of postpolypectomy bleeding for the large pedunculated colonic polyps.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pedunculated colorectal polyps, the heads of which were larger than 10mm and the stalk of which were large than 5 mm in diameter, were included.

Exclusion Criteria:

* bleeding tendency
* poor preparation
* sessile polyp

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Postpolypectomy bleeding | Immediate (bleeding occurring immediately after polypectomy and lasting for 30 s or more) and delayed bleeding complications were assessed. Delayed bleeding was subdivide into early (<24 h) and late (>24 h-30 days).

REFERENCES:
- [Derived] Ji JS, Lee SW, Kim TH, Cho YS, Kim HK, Lee KM, Kim SW, Choi H. Comparison of prophylactic clip and endoloop application for the prevention of postpolypectomy bleeding in pedunculated colonic polyps: a prospective, randomized, multicenter study. Endoscopy. 2014 Jul;46(7):598-604. doi: 10.1055/s-0034-1365515. Epub 2014 May 15. PMID 24830400